CLINICAL TRIAL: NCT06761482
Title: Non-Invasive Monitoring of Pediatric Kidney Transplant Recipients and Immunosuppression Personalization: an Open-labeled Multicenter Randomized Controlled Study
Acronym: MONITOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230817; IDRCB 2024-A01418-39 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-12-06; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Kidney Disease; Transplant;Failure,Kidney
Keywords: kidney; transplant; pediatric; rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: An open label multicenter prospective randomized trial of superiority with two active comparators / 4 groupes : monitoring by dd-cfDNA; monitoring by T-Vis; monitoring by dd-cfDNA+ T-Vis; Current standard of care based on surveillance biopsies and biological monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- monitoring by dd-cfDNA (Experimental)
  Interventions: Procedure: monitoring by dd-cfDNA
- monitoring by T-Vis (Experimental)
  Interventions: Procedure: monitoring by T-Vis
- monitoring by dd-cfDNA and T-Vis (Experimental)
  Interventions: Procedure: monitoring by dd-cfDNA+ T-Vis
- Current standard of care based on surveillance biopsies and biological monitoring (No Intervention)

INTERVENTIONS:
Procedure: monitoring by dd-cfDNA — monitoring by dd-cfDNA
  Arms: monitoring by dd-cfDNA
Procedure: monitoring by T-Vis — monitoring by T-Vis
  Arms: monitoring by T-Vis
Procedure: monitoring by dd-cfDNA+ T-Vis — monitoring by dd-cfDNA+ T-Vis
  Arms: monitoring by dd-cfDNA and T-Vis

SUMMARY:
Currently, the monitoring of children receiving a kidney transplantation includes surveillance biopsies to detect subclinical rejection and signs of toxicity of immunosuppressive drugs (tacrolimus).

The hypothesis of the study is that the combination of non-invasive biomarkers (Donor-derived cell-free DNA and Virus-specific T cells) will allow both the safe discontinuation of surveillance biopsies and the personalization of the exposure to calcineurin inhibitors among pediatric kidney transplant recipients.

DETAILED DESCRIPTION:
MONITOR is an open label multicenter prospective randomized trial of superiority with two active comparators (4 parallel groups 1:1:1:1).

Arm A: monitoring by dd-cfDNA; Arm B: monitoring by T-Vis; Arm C: monitoring by dd-cfDNA+ T-Vis; Comparator arm: Current standard of care based on surveillance biopsies and biological monitoring

Main objectives and primary endpoints :

1. To demonstrate that the use of an integrative score of allograft rejection including dd-cfDNA measurement allows the reduction of the number of surveillance biopsies.

   Endpoint: Number of biopsy performed in each arm
2. To demonstrate that steering immunosuppression based on Tvis numbers allows the reduction of the exposition to calcineurin inhibitors.

Endpoint: Tacrolimus exposure assessed as the mean of the residual concentration of Tacrolimus between M6 and M24

ELIGIBILITY:
Inclusion Criteria:

* Age less than 21 years old at transplantation
* Single renal transplant from a deceased or a living donor.
* Absence of pregnancy confirmed by a negative pregnancy test in women in child-bearing period.
* Subject and legal guardians are willing and able to provide signed written informed consent and to comply with the study procedures
* Patients affiliated to health insurance system including Aide Médicale de l'Etat (AME)

Exclusion Criteria:

* History of multi-organ transplant (interference with rejection natural history)
* No surveillance biopsy planned
* Adult patient (or legal guardians) with limited understanding of the French language preventing him from receiving informed information on the protocol

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of kidney allograft during the 2 years post-transplantation | 24 months
  To demonstrate that the use of an integrative score of allograft rejection including dd-cfDNA measurement allows the reduction of the number of surveillance biopsies.
Exposure to calcineurin inhibitors (mean tacrolimus level) between month 6 and month 24 post-transplantation. | 24 months
  To demonstrate that steering immunosuppression based on Tvis numbers allows the reduction of the exposition to calcineurin inhibitors.

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v4.0 in each group | 24 months
  Adverse events of particular interest will include de novo donor specific antibodies (DSA) formation, clinical rejection, plasma viral replication Cytomegalovirus Virus, Epstein-Barr virus, BK virus.
Cost-utility | 24 months
  Data sources for the latter will include the trial's case report form data for efficacy and resource consumption in terms of ambulatory care, informal care, and productivity losses. It will be complemented by participating hospitals' discharge data to gather information relative to hospital care and its associated costs. The effectiveness criteria will be the number of quality-adjusted life-years (QALYs) gained. QALYs will be derived from patients' responses to the EQ-5D questionnaire
Allograft fibrosis on the surveillance biopsy at 24 months | 24 months
Allograft function (estimated Glomerular Filtration Rate) at 24 months | 24 months
Predicted allograft survival until 10 years after evaluation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Julien HOGAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France